CLINICAL TRIAL: NCT06264570
Title: Evaluation of a Genetically Determined Personalized Approach in Prescribing Biologically Active Substances in Patients With Elevated Blood Homocysteine Levels, Prospective,Double-blind Randomised Trial.
Brief Title: Evaluation of a Genetically Determined Personalized Approach in Prescribing Biologically Active Substances in Patients With Elevated Blood Homocysteine Levels.
Acronym: PERBIO-HC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW007
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-03

CONDITIONS: Hyperhomocysteinemia
Keywords: Hyperhomocysteinemia; Cardiovascular diseases; Bioactive substances; Genetically-determined approach; Nutrigenomics
MeSH Terms: conditions — Hyperhomocysteinemia; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- B-TMG experimental group (Experimental): Subjects with normal COMT gene and MTHFR gene polymorphism
  Interventions: Dietary Supplement: B-TMG supplementation
- B-SAM experimental group (Experimental): Subjects with COMT gene polymorphism or normal COMT gene and normal MTHFR gene
  Interventions: Dietary Supplement: B-SAM supplementation
- B-TMG placebo group (Placebo Comparator): Subjects with normal COMT gene and MTHFR gene polymorph polymorphism ysm
  Interventions: Other: B-TMG placebo
- B-SAM placebo group (Placebo Comparator): Subjects with COMT gene polymorphism or normal COMT gene and normal MTHFR gene
  Interventions: Other: B-SAM placebo

INTERVENTIONS:
Dietary Supplement: B-TMG supplementation — B-TMG supplement (B2 riboflavin, B6 pyroxidine, B9 methylfolate, B12 methylcobalamine, S-adenosylmethionine, Trimethylglycerol (TMG), zinc sulfate) for subjects with normal COMT gene and MTHFR gene polymorphism
  Arms: B-TMG experimental group
Dietary Supplement: B-SAM supplementation — B-SAM supplement (B2 riboflavin, B6 pyroxidine, B9 folic acid, B12 adenosylcobalamin, magnesium, S-adenosylmethionine) for Subjects with COMT gene polymorphism or normal COMT gene and normal MTHFR gene
  Arms: B-SAM experimental group
Other: B-TMG placebo — B-TMG placebo for subjects with normal COMT gene and MTHFR gene polymorphism
  Arms: B-TMG placebo group
Other: B-SAM placebo — B-SAM placebo for Subjects with COMT gene polymorphism or normal COMT gene and normal MTHFR gene
  Arms: B-SAM placebo group

SUMMARY:
The clinical trial assesses the effectiveness and safety of a genetically-determined personalized approach to prescribing bioactive substances in patients with elevated blood homocysteine levels. Hyperhomocysteinemia (HHcy) is a risk factor for cardiovascular diseases (CVD), potentially exacerbating the effects of arterial hypertension and high cholesterol levels, increasing the risks of heart disease, stroke, and venous thrombosis. The trial aims to reduce plasma homocysteine levels to normal values (<15 µmol/L) through a pilot, single-center, prospective, double-blind, placebo-controlled study. The study will involve a 6-month observation period with visits at 1, 3, and 6 months, assessing the efficacy of two composite bioactive substances not considered medicinal drugs. The primary endpoint is the reduction of homocysteine levels in patients with elevated levels, while secondary endpoints include lowering very low-density lipoprotein levels, absence of anxiety and depression (using the Spielberg Anxiety Scale), and the occurrence of major cardiovascular events. The sample size is planned for 111 patients across three groups, with a 1:1:2 distribution, considering a 40% reduction in homocysteine levels in the treated group and 5% in the control group, aiming for an 80% power and a 0.05 alpha. Inclusion criteria include adults aged 18-80 with elevated homocysteine (>15 µmol/L) and LDL cholesterol levels (≥1.4 mmol/L), without taking any substances that could influence homocysteine levels for at least one month prior. The trial will also conduct an interim analysis after enrolling 55 patients, using statistical analysis to evaluate the results.

ELIGIBILITY:
Inclusion Criteria:

* Increased homocysteine level above 15 µmol/l;
* Increased LDL level >=1.4 mmol/l.;
* Absence of taking medications or any other products that may affect homocysteine levels in the blood for at least 1 month before enrollment in the study;

Exclusion Criteria:

* Individual intolerance to the components of the substance;
* Pregnancy or breastfeeding;
* Severe concomitant disease requiring constant monitoring (estimated survival less than 1 year);
* Taking dietary supplements or medications containing one of the components: dietary supplements for at least 3 months before inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in homocysteine levels in patients with elevated homocysteine levels in the blood evaluated by 15 µmol/l. | 6 months

SECONDARY OUTCOMES:
change in the level of very low density lipoproteins | 6 months
change of anxiety when using dietary supplements accessed by the Spielberg scale | 6 months
change of depression when using dietary supplements by the Becks scale | 6 months
occurrence of major cardiovascular events during follow-up | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia